CLINICAL TRIAL: NCT05139771
Title: An Open-label Multicenter Phase 2 Clinical Safety Investigation of the EndoArt® Implantation in Subjects With Chronic Corneal Edema
Brief Title: EndoArt® Implantation in Subjects With Chronic Corneal Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye-yon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLI-E033
Record Dates: First submitted 2021-10-20; First posted 2021-12-01 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2023-02

CONDITIONS: Corneal Edema
Keywords: Corneal edema; Chronic corneal edema; THE ENDOART®; Artificial Endothelial layer
MeSH Terms: conditions — Corneal Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoArt® Artificial Endothelial Layer (Other): EndoArt® is intended to be used as an endothelial prosthesis in patients with chronic corneal edema. One arm - all subjects will be implanted with EndoArt®.
  Interventions: Device: THE ENDOART® IMPLANTATION (Artificial Endothelial layer)

INTERVENTIONS:
Device: THE ENDOART® IMPLANTATION (Artificial Endothelial layer) — Implantation of EndoArt® is similar to other anterior segment surgical procedures such as DSAEK/DMEK.
  Other Names: DSAEK; DMEK

SUMMARY:
The EndoArt® is intended to be used as an endothelial prosthesis in patients with chronic corneal edema.The EndoArt® (Artificial Endothelial layer) is a permanent implant, constructed of a clear, transparent, foldable, biologically compatible copolymer of hydroxyethyl methacrylate and methyl methacrylate. The peripheral surface of the EndoArt® has either one or more marks, to ensure the correct orientation of the implant. The device serves as a physical barrier blocking the influx of water from the AC of the eye into the cornea due to dysfunctional corneal endothelial layer. Together with evaporation from the anterior surface of the cornea it maintains corneal hydration and clarity.

The EndoArt® device is CE marked approved (approved for marketing by the European regulatory authority).

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, phase 2 clinical investigation assessing safety of EndoArt® implantation, in subjects with chronic corneal edema. Safety will be assessed by evaluating the rate of adverse events and adverse device effects throughout the study period. Exploratory efficacy endpoints will be assessed by measuring the change in corneal thickness from baseline, change in pain score from baseline and changes in visual acuity. Time to, and rate of, post-surgical rebubbling to facilitate adhesion of the device will be explored.

Subjects with chronic corneal edema that meet the inclusion/exclusion criteria will be the study target population. The study will encompass a total of up to 80 subjects who will complete the Protocol follow-up schedule. For the Primary endpoint, the frequency and severity of device related adverse events, from patient entry through the 6-month follow-up period will be analyzed. Adverse events will be assessed on a continuous basis and will continue to be collected for 12 months.

This clinical investigation is conducted in up to 12 (twelve) clinical sites in Europe (Germany, France, and Netherlands), Mexico, India and Israel. Additional sites may be considered.

This clinical investigation has been designed to provide continuous clinical evidence for the EndoArt® as part of its clinical follow up program.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet the following inclusion criteria at screening visit:

1. Male or Female subjects 40-85 years of age.
2. Have chronic corneal edema (for a minimum of 3 months) secondary to endothelial dysfunction.
3. Have corneal thickness >600μm by OCT.
4. Have best corrected distance visual acuity 6/19 (20/63) or worse (equivalent ETDRS= 60 letters) with subjective symptoms of impaired visual function.
5. Subject with posterior pseudophakia and stable IOL.
6. Willing and able to understand and sign informed consent prior to any study related procedure.
7. Willing and able to follow study instructions (e.g., to lay on one's back for 4 hours post op), able to self-administer or have caregiver available to administer eyedrops as required by the protocol for the duration of the study, and able to attend study visits/assessments for the duration of the study.

Exclusion Criteria:

Individuals for participation will be ineligible for the study if any of the following conditions apply:

1. History of ocular Herpetic keratitis.
2. Scarred cornea resulting in visual impairment with intact endothelium (cell density ≥ 1500).
3. History of posterior vitrectomy.
4. Post PKP
5. Have an irregular posterior cornea (e.g., post trauma).
6. Have a current infection of the cornea.
7. Have band keratopathy and/or limbal stem cell deficiency.
8. Have clinically severe dry eye disease which needs more than 4 drops of lubricant per day.
9. Phthisis bulbi or subject is at risk of developing phthisis.
10. Subject with medically uncontrolled high intra ocular pressure.
11. Aphakia.
12. Anterior chamber IOL or fixated anterior chamber IOL.
13. Pseudophakodonesis.
14. Have large iris defect which could compromise intraoperative air bubble formation
15. Have undergone corneal refractive surgery.
16. History of neurotrophic cornea.
17. History of recurrent corneal erosion or persistent epithelial defect.
18. IridoCorneal Endothelial (ICE) Syndrome or any rare disease/ syndrome creating anatomical or physiological anomalies of the anterior chamber (e.g., corectopia).
19. Recurrent posterior, intermediate or anterior uveitis.
20. Subject receiving regular intravitreal injection
21. Currently participating or have participated in an investigational study, other than this study, within the past 60 days.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The frequency of device related adverse events (safety) | 12 months
  Adverse events will be assessed on a continuous basis from baseline until follow-ups completion.
The severity of device related adverse events (safety). | 12 months
  Adverse events will be assessed on a continuous basis from baseline until follow-ups completion.

SECONDARY OUTCOMES:
Change from baseline in central corneal thickness (CCT) postoperatively. | 6 months
  Central Corneal Thickness (pachymetry) will be measured by anterior segment Optical Coherence Tomography (OCT).
Incidence of primary post-surgical detachment of the device. | 12 months
  Post implantation device detachment
Rate of rebubbling post-op. | 12 months
  Number of times that post implantation re-bubbling is done
Change in Best Corrected Distance Visual Acuity (BCDVA) from baseline. | 12 months
  Visual acuity will be measured with ETDRS format charts.
Change in ocular pain score as assessed by a Visual Analogue Scale (VAS) from baseline. | 12 months
  VAS is a horizontal line, 0-100 mm. VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the subject marks.

CONTACTS AND LOCATIONS:
Locations (12):
- France (2):
  - Centre Hospitalier Régional Universitaire de Brest (CHRU Brest), Brest
  - Hôpital Fondation A. de Rothschild, Paris
- Georgia (4):
  - Akhali Mzera Eye Clinic, Tbilisi
  - Caucasus Medical Center (CMC), Tbilisi
  - Davinci Eye Medical Center, Tbilisi
  - High Technology Medical Center, University Clinic, Tbilisi
- International Vision Correction Research Centre (IVCRC) Universitätsklinikum Heidelberg, Heidelberg, Germany
- India (2):
  - Dr Agarwal's Eye Hospital, Tirunelveli, Tamil Nadu
  - L V Prasad Eye Institute, Hyderabad, Telangana
- Israel (2):
  - Rambam Medical Center, Haifa
  - Assuta HaShalom, Tel Aviv
- Amsterdam MC (AMC), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No